CLINICAL TRIAL: NCT03056833
Title: Phase I Trial of Ribociclib (Ribociclib (LEE-011)) With Platinum-based Chemotherapy in Recurrent Platinum Sensitive Ovarian Cancer
Brief Title: Ribociclib (Ribociclib (LEE-011)) With Platinum-based Chemotherapy in Recurrent Platinum Sensitive Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ronald Buckanovich (Other)
Responsible Party: Sponsor-Investigator, Ronald Buckanovich, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-006; CLEE011XUS28T (Other: Novartis, Inc)
Record Dates: First submitted 2017-02-14; First posted 2017-02-17 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-08

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — ribociclib; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ribociclib (Experimental): Ribociclib (LEE-011) will be used as concurrent therapy with platinum-based chemotherapy in platinum-sensitive recurrent ovarian cancer. Participants will receive 200, 400, or 600mg of ribociclib per day in combination with carboplatin + paclitaxel. Subjects will receive 6 cycles of carboplatin + paclitaxel given weekly with ribociclib.
  Interventions: Drug: ribociclib; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: ribociclib — Ribociclib (LEE-011) will be given on days 1-4, 8-11, and 15-18 of a 28 day cycle at 200, 400, or 600mg/day during the dose escalation phase. During the maintenance phase, ribociclib (LEE-011) will be given at 600mg/day, 3 weeks on, 1 week off until progression.
Drug: Paclitaxel — During the escalation phase Paclitaxel will be given on days 1, 8, and 15 of a 28 day cycle.
Drug: Carboplatin — During the escalation phase Carboplatin will be given on days 1, 8, and 15 of a 28 day cycle.

SUMMARY:
Investigators hypothesize that concurrent ribociclib treatment and chemotherapy will enhance the response to platinum-based therapy and maintenance therapy will slow ovarian cancer tumor growth leading to prolongation in progression free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 years old with platinum-sensitive recurrent ovarian, fallopian or primary peritoneal cancer (defined as recurrent disease >6 months after completing last platinum-based chemotherapy) eligible to receive platinum-based doublet chemotherapy.
2. Must have had at least 1 prior line of platinum-based therapy
3. ECOG 0-1 with life expectancy of ≥ 3 months
4. Adequate organ function:

   * Serum creatinine ≤1.5mg/dL or 24-hour clearance ≥50 mL/min
   * AST/ALT <2.5x ULN (or <5x ULN if liver metastasis are present)
   * Total bilirubin ≤ULN or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.
   * Hemoglobin ≥9 gm/dl, Platelets ≥100,000/µL, ANC ≥1500/µL
   * INR ≤1.5
   * Potassium, total calcium (corrected for serum albumin), magnesium, and sodium within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
5. Screening ECG (defined as the mean of the triplicate ECGs) with QTcF interval at screening ≤450msec (using Fridericia's correction) and resting heart rate 50-90bpm
6. Must be able to swallow ribociclib (LEE-011) tablet/capsule
7. Documented disease recurrence/progression based on GCIG-RECIST
8. Able to provide informed consent and comply with all study protocols
9. Treated CNS metastasis allowed if treatment is complete ≥8 weeks prior to enrollment. Patients must be asymptomatic off systemic corticosteroids for at least 4 weeks after completion of radiation therapy. CNS disease must be stable or regressed on repeat imaging performed at least 4 weeks after completion of therapy.
10. Women of child-bearing potential (those who have had a menstrual cycle within the last year and have not had a tubal ligation or surgical removal of both ovaries and/or hysterectomy) must agree to abstain from vaginal intercourse or use and continue highly effective methods of contraception for 3 weeks after discontinuation of study treatment.
11. Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.

Exclusion Criteria:

1. Borderline or low-malignant potential histology.
2. Platinum-resistant disease (as defined as progressive disease within 6 months of completion of chemotherapy with a platinum agent)
3. Grade 3 baseline neuropathy.
4. Known hypersensitivity to any of the excipients of ribociclib (LEE-011), including peanuts and soy
5. Prior use of CDK4/6 inhibitors.
6. Congenital long QT syndrome or family history of unexpected sudden cardiac death
7. Concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer or per physician discretion that the previous cancer was adequately treated with curative intent and unlikely to recur (the study PI must concur with this determination).
8. Impairment of gastrointestinal (GI) function or disease that may significantly alter the absorption of the study drugs
9. History of HIV infection
10. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks and contraindicate patient's participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
11. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

    a. Heart Association functional classification III-IV) b. Documented cardiomyopathy c. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening d. Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block) e. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following: i. Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesaemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.

    ii. Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication iii. Inability to determine the QT interval on screening (QTcF using Fridericia's correction) f. Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening g. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
12. Use of prohibited medications (see section 5.3) that cannot be changed to an alternative therapy
13. Patient is currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.

    a. The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
14. Patient is currently receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
15. Use of herbal supplements unless discontinued ≥7 days prior to initiation of study drug
16. Consumption of foods which are strong inducers or inhibitors of CYP3A4/5 has to be discontinued 7 days prior to initiation of study drug
17. Pregnancy or lactation
18. Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
19. Patient who has received radiotherapy ≤4 weeks or limited field radiation for palliation ≤2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥25% of the bone marrow (Ellis, 1961) was irradiated.
20. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
21. Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 5 Grade ≤1 (Exception to this criterion: patients with any grade of alopecia and/or neuropathy ≤ grade 2 are allowed to enter the study).
22. Patient with a Child-Pugh score B or C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women ≥18 years old
Enrollment: 35 (Actual)
Dates: Start 2017-06-10 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) of ribociclib (LEE-011) when given with carboplatin + paclitaxel in platinum-sensitive recurrent ovarian cancer | 56 days
  Participants will be observed for the first two treatment cycles (2, 28 day cycles) and maximum tolerated dose will be determined.

SECONDARY OUTCOMES:
Number of participants that respond to treatment | 18 months post treatment
  Overall response rate (ORR) will be analyzed. The number of patients that respond to treatment (exhibit Partial Response (PR) or Complete Response (CR)) will be recorded. PR is defined as at least a 50% reduction in CA 125 levels (response must be confirmed and maintained for at least 28 days) and/or at least 30% decrease in the sum diameters of target lesions. CR is defined as normalization of CA125 levels ((response must be confirmed and maintained for at least 28 days) and disappearance of all target lesions.
Time from treatment until disease progression or death | 18 months post treatment
  Progression is defined as one of the following:
  * Patients with elevated CA-125 pretreatment and normalization of CA-125 must show evidence of CA-125 greater than, or equal to, 2 times the upper limit of the reference range on 2 occasions at least 1 week apart or
  * Patients with elevated CA-125 before treatment, which never normalizes, must show evidence of CA-125 greater than, or equal to, 2 times the nadir value on 2 occasions at least 1 week apart or
  * Patients with CA-125 in the reference range before treatment must show evidence of CA-125 greater than, or equal to, 2 times the upper limit of the reference range on 2 occasions at least 1 week apart
  * Increase in at least 20% in sum of diameters of target lesions or any new lesions or unequivocal increase in non-target lesions.
  * Response determined via measurable disease (measurement of target and non-target lesions) takes precedence over CA125 criteria Stable Disease (SD): CA
Number of participants encountering toxicity at each dose level | 30 days post treatment
  Patients will potentially be treated with 3 different dose levels of ribociclib in combination with platinum-based chemotherapy.
Overall Survival (OS) | Up to 5 years
  The (median) length of time from start of treatment patients are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Lan G Coffman, M.D., Principal Investigator — University of Pittsburgh Medical Center
Locations (8):
- United States (8):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - UPMC Hillman Cancer Center Upper St. Clair, Bethel Park, Pennsylvania
  - UPMC Hillman Cancer Center Arnold Palmer at Mountain View, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center Arnold Palmer Medical at Norwin, Irwin, Pennsylvania
  - UPMC Hillman Cancer Center Arnold Palmer at Mt Pleasant, Mount Pleasant, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Passavant (OHA), Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center Washington, Washington, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coffman LG, Orellana TJ, Liu T, Frisbie LG, Normolle D, Griffith K, Uppal S, McLean K, Berger J, Boisen M, Courtney-Brooks M, Edwards RP, Lesnock J, Mahdi H, Olawaiye A, Sukumvanich P, Taylor SE, Buckanovich R. Phase I trial of ribociclib with platinum chemotherapy in ovarian cancer. JCI Insight. 2022 Sep 22;7(18):e160573. doi: 10.1172/jci.insight.160573. PMID 35972817